CLINICAL TRIAL: NCT05407142
Title: An Open Comprative Study of the Prophylactic Efficacy and a Non-comparative Study of the Immunogenicity and Safety of the Inactivated Whole-virion Concentrated Purified Coronavirus Vaccine (CoviVac), Produced by FSBSI "Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products", on Volunteers at the Age of 18-60 Years (Clinical Trials, Phase III)
Brief Title: An Open Comprative Study of the Prophylactic Efficacy and a Non-comparative Study of the Immunogenicity and Safety of the Inactivated Whole-virion Concentrated Purified Coronavirus Vaccine (CoviVac)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: № VKI-III-04/21
Record Dates: First submitted 2022-05-24; First posted 2022-06-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Coronavirus Infections; Vaccine
Keywords: COVID-19; Coronavirus infections; Vaccine; SARS-Cov-2; Immunobiological medicine
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The study group consisted of 3,500 volunteers who received the CoviVac vaccine (Experimental): Subgroup 1 - 2100 volunteers who will be vaccinated with the Nobivac vaccine twice with an interval of 21 days and revaccinated at 6 months with one dose of the KoviVac vaccine.
  Cohort 1 - The first 1000 volunteers of the study group will be used to assess the efficacy + safety + immunogenicity of the vaccine under study.
  Cohort 2 - Next 1100 volunteers of the study group will be used to analyze the efficacy + safety of the vaccine under study.
  Subgroup 2 - 1400 volunteers who will be vaccinated with CoviVac vaccine three times at intervals of 21 days intramuscularly at a dose of 0.5 ml.
  The data of 1400 volunteers vaccinated three times with an interval of 21 days will be used to assess the effectiveness + safety + immunogenicity of the vaccine under study.
  Interventions: Biological: CoviVac vaccine (inactivated whole-virion concentrated purified) manufactured by FSBSI "Chumakov FSC R&D IBP RAS"
- Control group (Other): The data from volunteers from the control group will be used to evaluate the effectiveness of the investigational vaccine.
  Interventions: Other: The data from volunteers from the control group

INTERVENTIONS:
Biological: CoviVac vaccine (inactivated whole-virion concentrated purified) manufactured by FSBSI "Chumakov FSC R&D IBP RAS" — Subgroup 1 - 2100 volunteers who will be vaccinated with the Nobivac vaccine twice with an interval of 21 days intramuscularly at a dose of 0.5 ml and revaccinated at 6 months with one dose of the KoviVac vaccine (0.5 ml).
  Subgroup 2 - 1400 volunteers who will be vaccinated with CoviVac vaccine three times at intervals of 21 days intramuscularly at a dose of 0.5 ml.
  Arms: The study group consisted of 3,500 volunteers who received the CoviVac vaccine
Other: The data from volunteers from the control group — Official data on the number of Covid-19 cases during the study period among 3,500 unvaccinated individuals.
  Arms: Control group

SUMMARY:
An Open Comprative Study of the Prophylactic Efficacy and a Non-comparative Study of the Immunogenicity and Safety of the Inactivated Whole-virion Concentrated Purified Coronavirus Vaccine (CoviVac), Produced by FSBSI "Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products", on Volunteers at the Age of 18-60 Years

DETAILED DESCRIPTION:
The study group is planned to screen a maximum of 32,000 volunteers inclusive, of which it is planned to include 3,500 men and women aged 18 to 60 years who meet the criteria for inclusion in the study and do not have non-inclusion criteria.

The study group consisted of 3,500 volunteers who received the CoviVac vaccine

Subgroup 1 - 2100 volunteers who will be vaccinated with the Nobivac vaccine twice with an interval of 21 days intramuscularly at a dose of 0.5 ml and revaccinated at 6 months with one dose of the KoviVac vaccine (0.5 ml).

Cohorts:

1. The data of the first 1000 volunteers of subgroup 1 will be used to assess the efficacy + safety + immunogenicity of the vaccine under study.
2. The data of the next 1100 volunteers of subgroup 1 will be used to analyze the efficacy + safety of the vaccine under study.

Subgroup 2 - 1400 volunteers who will be vaccinated with CoviVac vaccine three times at intervals of 21 days intramuscularly at a dose of 0.5 ml.

The data of 1400 volunteers vaccinated three times with an interval of 21 days will be used to assess the effectiveness + safety + immunogenicity of the vaccine under study

Control group - official data on the number of Covid-19 cases during the study period among 3,500 unvaccinated individuals.

The data of the control group volunteers will be used to evaluate the effectiveness of the vaccine under study.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must meet the following inclusion criteria:

Type of participants * Healthy volunteers or volunteers with a history of stable diseases that do not meet any of the criteria for non-inclusion in the study.

Age at the time of signing the Informed Consent * from ≥ 18 to < 60 years.

Paul * Male or female.

The volunteers of the study group must meet the following additional inclusion criteria:

* Written Informed consent of volunteers to participate in a clinical trial.
* Volunteers who are able to fulfill Protocol requirements (i.e. answer phone calls, fill out a Self-observation Diary, come to control visits).

  * For women capable of childbirth - a negative pregnancy test and consent to adhere to adequate methods of contraception (use of contraceptives within a month after the second vaccination). Women should use methods of contraception with a reliability of more than 90% (cervical caps with spermicide, diaphragms with spermicide, condoms, intrauterine spirals), or be sterile, or in a postmenopausal state.
  * For men capable of conception - consent to adhere to adequate methods of contraception (use of contraceptives within a month after the second vaccination). Men and their sexual partners should use methods of contraception with a reliability of more than 90% (cervical caps with spermicide, diaphragms with spermicide, condoms, intrauterine spirals), or be sterile.

Exclusion Criteria:

* Volunteers cannot be included in the study if any of the following criteria are present:

SARS-CoV-2 infection

* A case of established COVID-19 disease confirmed by PCR and/or ELISA in the last 6 months.

Diseases or medical conditions

* Severe and/or uncontrolled diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, gastrointestinal tract, liver, kidneys, hematopoietic, immune systems.
* Is registered at the dispensary for tuberculosis, leukemia, oncological diseases, autoimmune diseases.

  • Any confirmed or suspected immunosuppressive or immunodeficiency condition in the anamnesis.
* Splenectomy in the anamnesis.
* Neutropenia (decrease in the absolute number of neutrophils less than 1000/mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin less than 80 g/l) according to anamnesis.
* Anorexia.

Prior or concomitant therapy

* Vaccination with any vaccine carried out within 30 days before vaccination / the first dose of the studied vaccine or planned administration within 30 days after vaccination / the last dose of the studied vaccine.
* Prior vaccination with an experimental or registered vaccine that may affect the interpretation of the study data (any coronavirus or SARS vaccines).
* Long-term use (more than 14 days) of immunosuppressants or other immunomodulatory drugs (immunoregulatory peptides, cytokines, interferons, immune system effector proteins (immunoglobulins), interferon inducers (cycloferon) during the six months preceding the study, according to anamnesis.
* Treatment with glucocorticosteroids (≥ 20 mg of prednisone, or an analog, for more than 15 days during the last month).
* Volunteers who received immunoglobulin preparations or blood transfusion during the last 3 months before the start of the study according to anamnesis.

Other non-inclusion criteria

* Pregnancy or breast-feeding. Participation in any other clinical trial within the last 3 months.

Volunteers of the study group cannot be included in the study if any of the following criteria are present:

Diseases or medical conditions

* Serious post-vaccination reaction (temperature above 40 C, hyperemia or edema more than 8 cm in diameter) or complication (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions, accompanied or not accompanied by a feverish state) to any previous vaccination.
* Burdened allergic history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum sickness in the anamnesis, hypersensitivity or allergic reactions to the introduction of any vaccines in the anamnesis, known allergic reactions to vaccine components, etc.)•
* Guillain-Barre syndrome (acute polyradiculitis) in the anamnesis.
* The axillary temperature at the time of vaccination is more than 37.0 ° C.
* Acute infectious diseases (recovery earlier than 4 weeks before vaccination) according to anamnesis.
* Donation of blood or plasma (in the amount of 450 ml or more) less than 2 months before inclusion in the study.

Exclusion criteria:

* Withdrawal of Informed consent by a volunteer;

  * The volunteer was included in violation of the inclusion/non-inclusion criteria of the Protocol;

  • Any condition of a volunteer that requires, in the reasoned opinion of a medical researcher, the withdrawal of a volunteer from the study;

  * The established fact of pregnancy before the second vaccination;

  * The volunteer refuses to cooperate or is undisciplined (for example, failure to attend a scheduled visit without warning the researcher and/or loss of communication with the volunteer), or dropped out of observation;

  * For administrative reasons (termination of the study by the Sponsor or regulatory authorities), as well as in case of gross violations of the Protocol that may affect the results of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29000 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
Efficasy assessment | 12 month
  The proportion of vaccinated volunteers who do not have laboratory and clinically confirmed COVID-19 disease within 12 months after the second vaccination for all volunteers

SECONDARY OUTCOMES:
Classification by severity of COVID-19 | 12 month
  The proportion of study subjects with mild, moderate, severe and extremely severe COVID-19 that developed within 12 months after receiving the second dose of the vaccine from the total number of vaccinated for all volunteers.
The proportion of study subjects who died | 12 month
  The proportion of study subjects who died as a result of COVID-19 out of the number of cases for all volunteers.
The duration of laboratory and clinically confirmed COVID-19 disease. | 12 month
  The duration of laboratory and clinically confirmed COVID-19 disease
The proportion of volunteers from the total number of vaccinated / revaccinated with an increase in the level of the immune response | 12 month
  The proportion of volunteers from the total number of vaccinated / revaccinated with an increase in the level of the immune response in the form of an increase in geometric titers of specific antibodies (SGT) in the neutralization reaction and ELISA reaction." Only in cohort 1 of subgroup 1and subgroup 2.
Titer of specific antibody titer ≥ 4 times baseline Specific antibody titer ≥ 4 times baseline | 12 month
  The proportion of volunteers from the total number of vaccinated / revaccinated with a level of seroconversion (titer of specific antibodies ≥ 4 times from the initial level) in the virus neutralization reaction and the ELISA reaction.
  Only in cohort 1 of subgroup 1 and subgroup 2.
The level of γ-IFN and the subpopulation composition of T-lymphocytes. | 12 month
  The level of γ-IFN and the subpopulation composition of T-lymphocytes. Only in cohort 1 of subgroup 1 and subgroup 2.
Safety assessment | 12 month
  Frequency of occurrence of serious adverse events during the study.
Safety assessment | 12 month
  Frequency of occurrence, type and association with vaccination of adverse events during the study.
Safety assessment | 12 month
  Cases of early termination of volunteers' participation in the study due to the development of frequency incidence of adverse /serious frequency of adverse events associated with the use of research drugs.

CONTACTS AND LOCATIONS:
Locations (10):
- Russia (10):
  - Federal State Budgetary Educational Institution of Higher Education Kirov State Medical University of the Ministry of Health of Russia, Kirov
  - RUSAL Medical Center LLC, Krasnoyarsk
  - FSBI NIIVS named after I.I. Mechniko, Moscow
  - GBUZ "State Design Bureau named after D.D. Pletnev DZM", Moscow
  - "Scientific Research Institute of Occupational Medicine named after Academician N.F. Izmerov" (FGBNU "Research Institute of MT"), Moscow
  - CHUZ "Clinical Hospital "Russian Railways-Medicine" named after N.A. Semashko", Moscow
  - Limited Liability Company "H-Clinic" (LLC "H-Clinic"), Moscow
  - JSC "Medical services" CDL named after N.A.Semashko, Moscow
  - FSBSI Chumakov FSC R&D IBP RAS, Moscow, Russia, 108819
  - Mmc Sogaz Llc, Saint Petersburg